CLINICAL TRIAL: NCT03150680
Title: Development of a Risk Prediction Algorithm Through the Investigation of Genetic Risk Factors and the Complexity of Coronary Artery Disease to Estimate Future Risk of Cardiovascular Events: Angiographic (SYNTAX Score), Clinical and Pharmacogenetic Analysis.
Acronym: GESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AHEPA University Hospital (Other)
Collaborators: LABNET IAE - Private Reference Diagnostic Laboratory (Unknown)
Responsible Party: Principal Investigator, Georgios Sianos, Associate Professor of Cardiology MD, PhD, FESC, AHEPA University Hospital
Other Study IDs: CIP_GESS_Trial_1.1
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease
Keywords: SYNTAX score; SNPs; Genetics; Pharmacogenetics; Genetic Risk Score; Precision Medicine
MeSH Terms: conditions — Coronary Artery Disease; Genetic Risk Score | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — DNA will be extracted from obtained subject blood samples at the AHEPA University General Hospital of Thessaloniki. DNAs will be labeled by anonymized subject ID # (de-identified), and shipped to LABNET IAE - Private Reference Diagnostic Laboratory for genotyping and genetic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SYNTAX score = 0: Patients with nonobstructive CAD (≤50 % diameter stenosis)
  Interventions: Genetic: SNPs associated with CAD, SNPs associated with pharmacological response to clopidogrel and statins
- 0 < SYNTAX score <23: Low SYNTAX group
  Interventions: Genetic: SNPs associated with CAD, SNPs associated with pharmacological response to clopidogrel and statins
- SYNTAX score >= 23: Intermediate-High SYNTAX group
  Interventions: Genetic: SNPs associated with CAD, SNPs associated with pharmacological response to clopidogrel and statins

INTERVENTIONS:
Genetic: SNPs associated with CAD, SNPs associated with pharmacological response to clopidogrel and statins — Genotyping will be carried out by Next-Generation Sequencing (NGS)
  Other Names: Clinical information; Laboratory data

SUMMARY:
The purpose of the research project is to investigate the potential association of 207 genetic polymorphisms with the complexity and the severity of coronary artery disease (SYNTAX score), along with the patients' response to clopidogrel and statin therapy. The aim of the study is to combine genetic, pharmacogenetic, clinical and laboratory data in order to create an algorithm (GEnetic Syntax Score-GESS) that will enable an individualized therapeutic patient approach.

DETAILED DESCRIPTION:
Regarding Greece, this is the first prospectively enrolling medical database of this magnitude. Clinical and genetic patient information are systematically collected in a fashion that will enable also future retrospective evaluation of clinical and genetic details from each patient. This study is a discrete arm of a series of research projects that focus on the development of personalized medical therapy and share a common purpose: predicting future risk of cardiovascular events, assessing the severity and complexity of coronary artery disease by incorporating genetic information into the SYNTAX score and providing personalized therapeutic guidance to patients. The ultimate goal of the study would be to identify, design and develop a panel of genetic markers that in combination with clinical and angiographic information will be a reliable tool for predicting cardiovascular risk for future adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients giving voluntary written consent to participate in the study
2. Male or female patients between 18 years to 90 years at entry
3. Patients without previous history of CAD
4. Patients who are admitted in the Department of Cardiology in the AHEPA University General Hospital of Thessaloniki and undergo coronary angiography for clinical purposes

Exclusion Criteria:

1. Patients < 18 years old and > 90 years old at time of coronary angiography
2. Patients with a previous history of CAD
3. Cardiac Arrest at admission
4. Patients with serious concurrent disease and life expectancy of < 1 year
5. Patients who refuse to give written consent for participation in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 years to 90 years at entry, of both genders, who are admitted in the Department of Cardiology in the AHEPA University General Hospital of Thessaloniki and undergo coronary angiography for clinical purposes will be studied. Patients with a previous history of coronary artery disease will be excluded. The study includes subjects who 1) have suspected CAD and undergo a scheduled diagnostic angiogram for clinical reasons, and 2) are hospitalized because of an acute coronary syndrome and thus undergo diagnostic angiography (without previous history of CAD).
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Relationship between genetic risk variants and the SYNTAX score | 12 months
  All-comers population

SECONDARY OUTCOMES:
MACCEs | 12 months
  Cardiovascular death, myocardial infarction, stent thrombosis, any re-intervention and stroke
Predictive value of combining a Genetic Risk Score, SYNTAX score and clinical variables for the prediction of 1-year MACCEs | 12 months
  A multilocus Genetic Risk Score will be calculated as the weighted sum of alleles of 207 single nucleotide polymorphisms previously associated with CAD [The investigators will construct a multilocus genetic risk score for each individual by summing the number of risk alleles (0/1/2) for each of the 207 SNPs weighted by their estimated effect sizes].
  SYNTAX score is a coronary lesion complexity scoring system and represented by a single number.
  Clinical variables include:
  1. Major CV risk factors as defined according to ESC Guidelines [as dichotomous variables-yes or no]
  2. Ankle-Brachial Index: a tool for diagnosing peripheral artery disease but also an indicator of systemic atherosclerosis [measurement according to ESC Guidelines-represented by a single number]
  3. Left Ventricular Ejection Fraction (LVEF%) using echocardiography.
Any BARC (Bleeding Academic Research Consortium) bleeding | 12 months
  Bleeding Academic Research Consortium (BARC) recently proposed a novel standardized bleeding definition

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Sianos, MD PhD FESC, Principal Investigator — AHEPA University Hospital
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Background] Vizirianakis IS. Challenges in current drug delivery from the potential application of pharmacogenomics and personalized medicine in clinical practice. Curr Drug Deliv. 2004 Jan;1(1):73-80. doi: 10.2174/1567201043480009. PMID 16305372
- [Derived] Vizirianakis IS, Chatzopoulou F, Papazoglou AS, Karagiannidis E, Sofidis G, Stalikas N, Stefopoulos C, Kyritsis KA, Mittas N, Theodoroula NF, Lampri A, Mezarli E, Kartas A, Chatzidimitriou D, Papa-Konidari A, Angelis E, Karvounis Eta, Sianos G. The GEnetic Syntax Score: a genetic risk assessment implementation tool grading the complexity of coronary artery disease-rationale and design of the GESS study. BMC Cardiovasc Disord. 2021 Jun 8;21(1):284. doi: 10.1186/s12872-021-02092-5. PMID 34103005